CLINICAL TRIAL: NCT01125280
Title: Prospective Multicenter Validation of a Clinicoradiological Score for Predicting the Severity of Strangulated Small Bowel Occlusion
Brief Title: Prospective Multicenter Validation of a Severity Score of Strangulated Small Bowel Occlusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Geneva (Other)
Collaborators: Centre Hospitalier Universitaire Vaudois (Other)
Responsible Party: Schwenter Frank, MD, PhD, Geneva University Hospital, Department of Surgery
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NAC 10-009
Record Dates: First submitted 2010-05-17; First posted 2010-05-18 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Intestinal Obstruction
Keywords: Small bowel occlusion; Conservative treatment for small bowel occlusion; Surgical treatment for small bowel occlusion; Small bowel resection; Score of severity of small bowel occlusion
MeSH Terms: conditions — Intestinal Obstruction | interventions — Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SBO score application (Experimental): Acute strangulated SBO patients will receive a severity score at emergency admission. According to the score, they will be managed either conservatively or surgically. During surgery, the need of small bowel resection will be evaluated. The endpoint will be to correlate the type and success of treatment with the score in order to validate this new tool in SBO assessment.
  Interventions: Procedure: Conservative treatment versus surgical treatment

INTERVENTIONS:
Procedure: Conservative treatment versus surgical treatment — Conservative treatment: starving, nasogastric tube Surgical treatment: open laparotomy, adhesiolysis, with or without small bowel resection
  Other Names: Laparotomy; Adhesiolysis; Small bowel resection

SUMMARY:
The purpose of this study is to apply and validate a clinicoradiological score for the prediction of severity of strangulated small bowel occlusion (SBO). This score was elaborated by analyzing clinical, biological and radiological parameters of patients admitted in an emergency center for acute strangulated SBO. Two clinical, two biological and two radiological parameters were shown to significantly predict the surgical outcome of SBO patients.

Since any delay in the management of SBO may result in devastating consequences, a score predicting the severity of the SBO episode is an essential tool for helping in the management of SBO patients. A prospective multicenter validation of the score is mandatory for its extended use.

DETAILED DESCRIPTION:
Elaboration of the SBO score:

Intestinal ischaemia as a result of small bowel obstruction (SBO) requires prompt recognition and early intervention. A clinicoradiological score was sought to predict the risk of ischaemia in patients with SBO. A determined protocol for the assessment of patients presenting with SBO was used. A logistic regression model was applied to identify determinant variables and construct a clinical score that would predict ischaemia requiring resection. Of 233 successive patients with SBO, 138 required laparotomy of whom 45 underwent intestinal resection. In multivariable analysis, six variables correlated with small bowel resection and were given one point each towards the clinical score: history of pain lasting more than 4 days, guarding, C-reactive protein level at least 75 mg/l, leucocyte count over 10 G/l, free intraperitoneal fluid volume exceeding 500 ml on computed tomography (CT) and reduction of CT small bowel wall contrast enhancement. The risk of intestinal ischaemia was 6 per cent in patients with a score of 1 or less, whereas 21 of 29 patients with a score of three or more 3 underwent small bowel resection. A positive score of 3 or more had a sensitivity of 67.7 per cent and specificity 90.8 per cent; the area under the receiver operating characteristics curve was 0.87 (95 per cent confidence interval 0.79 to 0.95). By combining clinical, laboratory and radiological parameters, the clinical score allowed early identification of strangulated SBO.

The purpose of the present protocol is to apply the SBO score as a prospective multicenter study. After informed consent, SBO patients corresponding to the inclusion and exclusion criteria will be managed according to the score. Patients with a score of 0 to 2 will be treated conservatively, while a score ≥3 will imply emergency surgery. For its validation, the conservative and surgical outcomes will be compared with the results obtained for the elaboration of the score.

ELIGIBILITY:
Inclusion Criteria:

* Strangulated small bowel occlusion
* Diagnosis confirmation by CT-scan with iv contrast
* Blood analysis comprising: leucocyte count and repartition, CRP, lactates

Exclusion Criteria:

* Large bowel occlusion
* Strangulated hernia
* Tumor occlusion
* Post-Radiotherapy occlusion
* Paralytic ileus (neurological diseases, diabetes, etc)
* Inflammatory bowel diseases
* Any condition able to modify the clinical or biological parameters without any relation with the SBO episode (inflammatory, infectious diseases, etc)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with a score of 0-2 with successful conservative treatment | 3 days
  According to the score, patients will be managed either conservatively or surgically. Patients with a score of 0-2 will be treated conservatively. The success of the decision and the treatment will be evaluated after 3 days since admission. Indeed, patients with conservative treatment who do not retrieve a gastrointestinal transit after 3 days will be operated on.

SECONDARY OUTCOMES:
Proportion of patients with a score ≥3 needing small bowel resection | 1 day
  Patients with a score ≥3 will be emergently operated on with a surgical delay below 12 hours since admission. During surgery, segmental small bowel resection will be performed in case of ischemia or necrosis. The need of small bowel resection will be related to the pre-operative score.

CONTACTS AND LOCATIONS:
Overall Officials: Frank P Schwenter, MD, PhD, Principal Investigator — University Hospital, Geneva
Locations (1):
- Division of visceral and transplantation surgery, Department of surgery, Geneva University Hospital, Geneva, Canton of Geneva, Switzerland

REFERENCES:
- [Derived] Wassmer CH, Revol R, Uhe I, Chevallay M, Toso C, Gervaz P, Morel P, Poletti PA, Platon A, Ris F, Schwenter F, Perneger T, Meier RPH. A new clinical severity score for the management of acute small bowel obstruction in predicting bowel ischemia: a cohort study. Int J Surg. 2023 Jun 1;109(6):1620-1628. doi: 10.1097/JS9.0000000000000171. PMID 37026805